CLINICAL TRIAL: NCT04782076
Title: An Open-Label Study to Investigate the Effect of Selpercatinib on the Pharmacokinetics of Dabigatran in Healthy Volunteers
Brief Title: A Drug Drug Interaction (DDI) Study of Selpercatinib and Dabigatran in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Loxo Oncology, Inc. (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 17972; J2G-MC-JZJV (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-03-02; First posted 2021-03-04 (Actual); Results first posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran; selpercatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dabigatran + Selpercatinib (Experimental): Participants received a single oral dose of 150 milligrams (mg) dabigatran on Day 1 and a single oral dose of 150 mg dabigatran coadministered with a single oral dose of 2 x 80 mg (160 mg) selpercatinib on Day 8.
  There was a washout period of 7 days between dosing on Days 1 and 8.
  Interventions: Drug: Dabigatran; Drug: Selpercatinib

INTERVENTIONS:
Drug: Dabigatran — Administered orally.
Drug: Selpercatinib — Administered orally.
  Other Names: LY3527723

SUMMARY:
The main purpose of this study is to determine the effect of selpercatinib on the levels of dabigatran in the blood stream and how long it takes the body to remove dabigatran. This study will also look at how safe and well-tolerated of dabigatran when administered in combination with selpercatinib in healthy participants. This study will last approximately 22 to 25 days.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males or females, as determined by medical history, physical examination and vital signs.
* Body mass index (BMI) within the range of 19 to 35 kilograms per meter squared (kg/m²)
* Male participants are not required to adhere to contraceptive requirements and female participants of childbearing potential must agree to be either remain abstinent or stay in a same sex relationship without sexual relationships with males or must agree to use a highly effective method of contraception and who underwent bilateral salpingectomy. The Female participants not of childbearing potential are not required to use contraception.

Exclusion Criteria:

* Have a positive pregnancy test at screening or Day -1, where applicable
* Are planning to become pregnant during the study or within 1 month of study completion
* Are women who are lactating
* Have known allergies to selpercatinib- or dabigatran-related compounds or any components of the formulation of selpercatinib or dabigatran, or history of significant atopy
* Have a history of allergic reactions to medications or food products
* Have a clinically significant abnormality of blood pressure and/or pulse rate as determined by the investigator
* Have known bleeding disorder including prior personal or familiar history of abnormal bleeding, hereditary or acquired coagulation or platelet disorder
* Clinically significant abnormalities on ECG as determined by the investigator or prolongation of the QTcB or QTcF >450 msec on more than 1 ECG obtained during screening only
* Have clinically significant active cardiovascular disease or history of myocardial infarction within 6 months prior to the planned start of selpercatinib
* Are currently enrolled in any other clinical study involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study
* Have an average weekly alcohol intake that exceeds 21 units per week (males ≤65 years old) and 14 units per week (females); 1 unit = 12 oz or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirit(s)
* Are smokers of more than 10 cigarettes or e-cigarettes, or 3 cigars or 3 pipes, per day
* Consume excessive amounts of coffee, tea, cola, or other caffeinated beverages per day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Inc, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dabigatran + Selpercatinib
Started | 36
Received at Least One Dose of Dabigatran on Day 1 | 36
Washout Period | 36
Received at Least One Dose of Selpercatinib and Dabigatran on Day 8 | 35
Completed | 35
Not Completed | 1
Not completed — Family Emergency | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Arm/Group | Dabigatran + Selpercatinib
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Dabigatran
Description: PK: Cmax of Dabigatran
Time Frame: Day 1 and Day 8: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hours (h) postdose
Population: All participants who received at least one dose of dabigatran and had evaluable PK.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Dabigatran: Participants received a single oral dose of 150 milligrams (mg) dabigatran on Day 1.
- Selpercatinib + Dabigatran: Participants received a single oral dose of 150 mg dabigatran coadministered with a single oral dose of 2 x 80 mg (160 mg) Selpercatinib on Day 8.
Arm/Group | Dabigatran | Selpercatinib + Dabigatran
Number analyzed (Participants) | 36 | 35
nanogram per milliliter (ng/mL) | 192 (41) | 276 (36)
Statistical Analysis 1: Comparison: Dabigatran vs Selpercatinib + Dabigatran; Test type: Other; Mixed Models Analysis; Least Squares Mean (LS Mean); LS Mean Difference (Final Values) = 1.43, 90% CI 2-sided [1.33 to 1.55]

2. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-inf]) of Dabigatran
Description: PK: AUC(0-inf) of Dabigatran
Time Frame: Day 1 and Day 8: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 h postdose
Population: All participants who received at least one dose of dabigatran had evaluable PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Dabigatran | Selpercatinib + Dabigatran
Number analyzed (Participants) | 36 | 35
nanogram*hour per milliliter (ng*h/mL) | 1650 (42) | 2290 (37)
Statistical Analysis 1: Comparison: Dabigatran vs Selpercatinib + Dabigatran; Test type: Other; Mixed Models Analysis; LS Mean Difference (Final Values) = 1.38, 90% CI 2-sided [1.30 to 1.46]

3. Secondary Outcome: PK: Cmax of Selpercatinib
Description: PK: Cmax of Selpercatinib
Time Frame: Day 8: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 h postdose
Population: All participants who received at least one dose of Selpercatinib and had evaluable PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Selpercatinib + Dabigatran
Number analyzed (Participants) | 35
ng/mL | 1830 (23)

4. Secondary Outcome: PK: AUC(0-inf) of Selpercatinib
Description: PK: AUC(0-inf) of Selpercatinib
Time Frame: Day 8: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 h postdose
Population: All participants who received at least one dose of Selpercatinib and had evaluable PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Selpercatinib + Dabigatran
Number analyzed (Participants) | 35
ng*h/mL | 25600 (27)

5. Secondary Outcome: PK: Time of Maximum Observed Drug Concentration (Tmax) of Selpercatinib
Description: PK: Tmax of Selpercatinib
Time Frame: Day 8: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 h postdose
Population: All participants who received at least one dose of Selpercatinib and had evaluable PK.
Measure: Median (Full Range); unit: hours
Arm/Group | Selpercatinib + Dabigatran
Number analyzed (Participants) | 35
hours | 3.00 [1.50 to 6.00]

ADVERSE EVENTS:
Time Frame: Baseline up to 25 days
Description: All participants who received at least one dose of study drug.
Groups:
- 150 mg Dabigatran: Participants received a single oral dose of 150 milligrams (mg) dabigatran on Day 1.
- 150 mg Dabigatran + 160 mg Selpercatinib: Participants received a single oral dose of 150 mg dabigatran coadministered with a single oral dose of 2 x 80 mg (160 mg) selpercatinib on Day 8.
Arm/Group | 150 mg Dabigatran | 150 mg Dabigatran + 160 mg Selpercatinib
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/35
Other Adverse Events (participants affected / at risk) | 0/36 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT04782076/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/76/NCT04782076/SAP_001.pdf